CLINICAL TRIAL: NCT00201799
Title: Phase II Trial of Infliximab for the Prevention of Acute Graft-versus-Host Disease Following Allogenic Hematopoietic Stem Cell Transplantation
Brief Title: Infliximab for the Prevention of Graft-versus-Host Disease Following Allogenic Hematopoietic Stem Cell Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Craig Hofmeister, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: OSU-0323
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2015-06-10 (Estimated); Status verified 2015-06

CONDITIONS: Graft-Versus-Host Disease
Keywords: Hematopoietic Stem Cell Transplantation
MeSH Terms: conditions — Graft vs Host Disease | interventions — Infliximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Infliximab (Experimental): Patients will be treated with infliximab day 1 prior to starting myeloblative chemotherapy or radiotherapy. A total of 6 doses will be administered.
  Interventions: Drug: Infliximab

INTERVENTIONS:
Drug: Infliximab — A total of 6 doses of Infliximab will be administered as follows:
  Dose 1: 10 mg/kg IV one day prior to commencing the myeloablative preparative regimen Dose 2: 10 mg/kg IV on day 0 to be given after peripheral blood stem cell infusion Dose 3: 10 mg/kg IV on day +7 Dose 4: 10 mg/kg IV on day +14 Dose 5: 10 mg/kg IV on day +28 Dose 6: 10 mg/kg IV on day +42
  Other Names: (Remicade®, Centocor)

SUMMARY:
This study will evaluate the efficacy of infliximab in reducing the incidence of grade II-IV acute graft versus host disease by day +100 post-transplant in patients undergoing allogeneic hematopoietic stem cell transplant.

DETAILED DESCRIPTION:
Rationale: Acute graft host disease (GvHD) remains a barrier to successful hematopoietic stem cell transplantation (HCT) used for the treatment of cancers in some patients. GvHD can result from a lack of compatibility between the donor and recipient. Research suggests another primary cause of GvHD comes from cytokines, or a substance produced by cells of the immune system that affect the immune response in both positive and negative ways. Infliximab is an antibody that directly targets the cytokine associated with GvHD. This study is building upon previous research to assess infliximab's ability to prevent GvHD after HCT.

Purpose: This study is evaluating the efficacy of infliximab in reducing the incidence of GvHD after HCT. The safety of this approach, along with changes to specific cytokines from this treatment, will also be measured.

Treatment: Patients in this study will receive infliximab through intravenous infusion. Infliximab will be administered in six doses, including one day before chemotherapy or radiotherapy, after the stem cell infusion, and then on days 7, 14, 28 and 42. Standard post-transplant treatments of cyclosporine (Neoral) and methotrexate (Methotrexate) will also be given through intravenous infusion. Cyclosporine will be given on day 1, and the subsequent schedule will be determined on an individual basis. Methotrexate will be administered on days 1, 3, 6, and 11. Several tests and exams will be given throughout the study to closely monitor patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing allogeneic HCT for the following disorders:

  * Acute myelogenous leukemia
  * Acute lymphoblastic leukemia
  * Non-Hodgkin's lymphoma
  * Hodgkin's disease
  * Multiple myeloma
  * Chronic lymphocytic leukemia
  * Chronic myeloid leukemia in accelerated or blast crisis at time of transplant.
* Age >20 yrs

Exclusion Criteria:

* Patients undergoing allogeneic stem cell transplantation for chronic myelogenous leukemia and aplastic anemia are excluded.
* Pregnant or breast-feeding females.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2004-02; Primary Completion 2006-08 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Evaluate efficacy of infliximab in reducing incidence of grade II-IV acute GvHD by day +100 post transplant in patients undergoing allogenic HCT and receiving standard cyclosporine and short course methotrexate GvHD prophylaxis. | 2004-2008
  * For matched related donor transplants, we will test the null hypothesis H0: p ≥0.40 versus the alternative H1: p≤0.20, where p is the probability of grade II-IV acute GvHD by day +100.
  * For matched unrelated donor transplants, we will test the null hypothesis H0: p≥0.70 versus the alternative H1: p≤0.50, where p is the probability of grade II-IV acute GvHD by day +100.

SECONDARY OUTCOMES:
Assess the effect of infliximab on treatment-related mortality at 100 days post-transplant and on the incidence and severity of regimen related toxicity, including veno-occlusive disease (VOD) of the liver and interstitial pneumonitis (IP). | 2004-2008
  * Describe the incidence of infections occurring during the first year post-transplant.
  * Assess the effect of infliximab on the incidence of chronic GvHD
  * Relapse rate of the primary hematological malignancy
  * Assess the effect of Infliximab on blocking the TNF response to the conditioning regimen, and on the changes in cytokines important in the pathogenesis of acute GvHD in the peritransplant setting.
  * Explore the relationship between TNF gene polymorphism on the efficacy of infliximab prophylaxis therapy in preventing acute GvHD.

CONTACTS AND LOCATIONS:
Overall Officials: Craig Hofmeister, MD, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University, Columbus, Ohio, United States

REFERENCES:
- [Result] Hamadani M, Hofmeister CC, Jansak B, Phillips G, Elder P, Blum W, Penza S, Lin TS, Klisovic R, Marcucci G, Farag SS, Devine SM. Addition of infliximab to standard acute graft-versus-host disease prophylaxis following allogeneic peripheral blood cell transplantation. Biol Blood Marrow Transplant. 2008 Jul;14(7):783-9. doi: 10.1016/j.bbmt.2008.04.006. PMID 18541197
- See also: Jamesline — http://cancer.osu.edu